CLINICAL TRIAL: NCT04097197
Title: Factors Influencing Flu Vaccination in Primary Health Care
Acronym: FIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agrupamento de Centros de Saúde de Dão Lafões (Other)
Responsible Party: Principal Investigator, Frederico Rosário, Head of Research Department, Agrupamento de Centros de Saúde de Dão Lafões
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIVA_2019
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Flu, Human
Keywords: Influenza Vaccines; Influenza, Human; Primary Health Care
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Before-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving information (Experimental): Patients in the experimental arm will receive a brief educational intervention if they initially refuse flu vaccination. The intervention was designed towards the most common barriers to flu vaccination that were found after a brief review of the literature. After the intervention, patients will be asked again whether or not they wish to receive the flu vaccine.
  Interventions: Behavioral: Brief educational intervention

INTERVENTIONS:
Behavioral: Brief educational intervention — same as before

SUMMARY:
This study aims to study the barriers to flu vaccination among at-risk people at the Primary Health Care level in order to increase the vaccination rates as recommended by the World Health Organization.

DETAILED DESCRIPTION:
People from vulnerable groups (e.g., those diagnosed with Diabetes, Chronic Obstructive Pulmonary Disease, Asthma) are at increased risk of developing complications from infection with influenza virus, that could ultimately result in death.

Flu vaccination is recommended by many authorities, including the World Health Organization, as a means to decrease the risk of developing such life-threatening conditions. However, vaccination rates are well below the recommended threshold.

ELIGIBILITY:
Inclusion Criteria:

* People 65+ otherwise healthy;
* Patients of any age diagnosed with at least one of the following conditions: Diabetes, Asthma, COPD, Coronary Disease or Hearth failure;
* No history of flu vaccination in the previous year.

Exclusion Criteria:

* Patients who have been vaccinated against the flu but who have no record of it in the clinical records;
* Patients with contraindications to flu vaccination;
* Patients that cannot be reached either by phone or letter.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Flu vaccination refusal rate | up to 6 months
  Percentage of patients refusing flu vaccination prior to intervention

SECONDARY OUTCOMES:
Prevalence of barriers to flu vaccination | up to 6 months
  Percentage of participants mentioning a determined barrier to flu vaccination
Flu vaccination acceptance rate post-intervention | up to 6 months
  Percentage of patients who accept receiving the flu vaccine after receiving the intervention
Flu vaccination rate | up to 6 months
  Percentage of patients who have been vaccinated after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Dão Lafões Grouping of Primary Health Care Centres, Viseu, Dão Lafões, Portugal

IPD SHARING:
Plan to Share IPD: No